CLINICAL TRIAL: NCT06165016
Title: Far Red Light to Improve Functioning in PAD: The LIGHT PAD Trial
Brief Title: Far Red Light to Improve Functioning in PAD
Acronym: LIGHT PAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Mary McDermott, Jeremiah Stamler Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00218660
Record Dates: First submitted 2023-11-19; First posted 2023-12-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Artery Disease; Peripheral Vascular Disease; Aging; Walking, Difficulty
Keywords: light therapy
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Investigators will randomize 32 participants age 50 and older with PAD to one of two groups: far red light therapy or sham therapy. Participants will be followed for four months.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This will be a double blinded study where both the participant and the people collecting data will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Far red light therapy (Experimental): Subgroup of participants receiving the 670 nm far red light device
  Interventions: Device: Far red light therapy
- Sham therapy (Sham Comparator): Subgroup of participants receiving the sham light device, far red light device covered with blue filter paper to block 670 nm light, resulting in mean power generated of 0.24 mW/cm2, compared to 26.3 mW/cm2 for the intervention, a 100-fold difference.
  Interventions: Device: Sham light therapy

INTERVENTIONS:
Device: Far red light therapy — All participants will receive one far red light device per leg. Participants will be asked to use their two light devices daily, exposing their bare legs to the devices for 10 minutes twice per day. A study coordinator will deliver the light devices to each participant's home, positioning the devices 15 cm behind the participant's heels, using tape on the floor to mark where the light and feet should be positioned. Twice each day, the participant flips a switch on the device to begin each session. A timer will turn off the device after 10 minutes. A power meter will measure the total time that the device was turned on. Participants will also record use of the light in a log.
  Arms: Far red light therapy
Device: Sham light therapy — All participants will receive one sham device per leg. Participants will be asked to use their two light devices daily, exposing their bare legs to the devices for 10 minutes twice per day. A study coordinator will deliver the light devices to each participant's home, positioning the devices 15 cm behind the participant's heels, using tape on the floor to mark where the light and feet should be positioned. Twice each day, the participant flips a switch on the device to begin each session. A timer will turn off the device after 10 minutes. A power meter will measure the total time that the device was turned on. Participants will also record use of the light in a log.
  Arms: Sham therapy

SUMMARY:
The LIGHT PAD Trial is a Phase II multi-centered randomized clinical trial to collect preliminary data to test whether daily far red light treatment of the lower extremities in people with PAD improves six-minute walk distance, lower extremity perfusion, and ischemia-related damage in gastrocnemius muscle at four-month follow-up, compared to a sham control. Participants will complete 10 minutes of twice daily home treatment with either far red light or a sham light for four months.

DETAILED DESCRIPTION:
The LIGHT PAD Trial is a Phase II multi-centered randomized clinical trial to collect preliminary data to test whether daily far red light treatment of the lower extremities in people with PAD improves six-minute walk distance, lower extremity perfusion, and ischemia-related damage in gastrocnemius muscle at four-month follow-up, compared to a sham control. Participants will complete 10 minutes of twice daily home treatment with either far red light or a sham light for four months.

Participants with PAD will be randomized at one of two centers: Northwestern University (PI: MM McDermott, MD) and the University of Alabama (PI: Nicole Lohr MD, PhD) to daily far red light or sham control for four months. The primary outcome, change in six-minute walk, will be measured at four month follow-up, immediately after the final administration of far red light or sham. In secondary and exploratory aims, investigators will distinguish between acute and chronic effects of far red light on six-minute walk, measure the effects of far red light on patient-reported outcomes, and delineate biologic pathways by which far red light improves walking performance in PAD, by measuring change in plasma nitrite and nitrosothiols, gastrocnemius muscle perfusion (MRI arterial spin labeling) and gastrocnemius muscle health and mitochondrial activity. If the proposed hypotheses are supported by this Phase II trial, results will be used to design a definitive randomized trial of far red light for people with PAD.

To achieve the specific aims, investigators will randomize 32 participants age 50 and older with PAD to one of two groups: far red light therapy or sham therapy. Participants will be followed for four months.

ELIGIBILITY:
Inclusion Criteria.

First, all participants will be age 50 and older. Second, all participants will have PAD. PAD will be defined as:

1. An ABI <= 0.90 at baseline.
2. Vascular lab evidence of PAD (such as a toe brachial pressure =< 0.70 or an ankle brachial index less than or equal to 0.90), or angiographic evidence of PAD defined as at least 70% stenosis of an artery supplying the lower extremities.
3. An ABI of >0.90 and <= 1.00 who experience a 20% or greater drop in ABI in either leg after the heel-rise test.

Exclusion Criteria:

1. Above- or below-knee amputation
2. Critical limb ischemia defined as an ABI <0.40 with symptoms of rest pain
3. Wheelchair confinement or requiring a walker to ambulate
4. Walking is limited by a symptom other than PAD
5. Current foot ulcer on bottom of foot
6. Failure to successfully complete the study run-in
7. Planned major surgery, coronary or leg revascularization during the next four months
8. Major surgery, coronary or leg revascularization or major cardiovascular event in the previous three months
9. Major medical illness including lung disease requiring oxygen, Parkinson's disease, a life-threatening illness with life expectancy less than six months, or cancer requiring treatment in the previous two years. [NOTE: potential participants may still qualify if they have had treatment for an early stage cancer in the past two years and the prognosis is excellent, unless the cancer is located in the lower extremities. Participants who require oxygen only at night may still qualify.]
10. Mini-Mental Status Examination (MMSE) score < 23
11. Non-English speaking
12. Participation in or completion of a clinical trial in the previous three months. [NOTE: after completing a stem cell or gene therapy intervention, participants will become eligible after the final study follow-up visit of the stem cell or gene therapy study so long as at least six months have passed since the final intervention administration. After completing a supplement or drug therapy (other than stem cell or gene therapy), participants will be eligible after the final study follow-up visit as long as at least three months have passed since the final intervention of the trial.]
13. Visual impairment that limits walking ability.
14. Six-minute walk distance of <400 feet or >1700 feet.
15. Participation in a supervised treadmill exercise program or a cardiac rehabilitation program in previous three months or planning to begin a supervised treadmill exercise program or a cardiac rehabilitation program in the next five months.
16. Unwilling to avoid red light therapy outside of study participation.
17. Baseline blood pressure <100/45.
18. In addition to the above criteria, investigator discretion will be used to determine if the trial is unsafe or not a good fit for the potential participant.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Walk Distance | Measured at baseline and 4 month follow-up
  Four month change in six-minute walk distance

SECONDARY OUTCOMES:
Walking Impairment Questionnaire Distance (WIQ) Score | Measured at baseline and 4 month follow-up
  Four month change in the WIQ distance score. Score range 0-100, 100 is best
Six-Minute Walk Distance | Measured immediately after the first light treatment (within 15 minutes after the first treatment, acute effect)
  Acute change in six-minute walk distance after first light therapy
Six-minute walk distance. | Measured at 4-month follow-up, 24 hours after the final treatment.
  Four month change in 6-minute walk, measured 24 hours after last treatment.
Calf muscle perfusion | Measured at baseline and four-month follow up
  Changes in calf muscle perfusion at 3 Tesla measured with arterial spin labeling with MRI and post-cuff occlusion hyperemia

OTHER OUTCOMES:
Plasma nitrite | Measured before and within five minutes after the first light treatment
  Acute change in plasma abundance of nitrite
Plasma nitrite | Measured before and within five minutes after the final light treatment at four-month follow up
  Four- month changes in plasma abundance of nitrite
Plasma Nitrosothiols | Measured before and within five minutes after the first light treatment
  Changes in plasma abundance of nitrosothiols
Plasma Nitrosothiols | Measured before and within five minutes after the final light treatment at four-month follow up.
  Changes in plasma abundance of nitrosothiols
Gastrocnemius Muscle Capillary Density | Measured at baseline and four-month follow up
  Four month changes in gastrocnemius muscle capillary density
Gastrocnemius Muscle Myofiber Size | Measured at baseline and four-month follow up
  Four month changes in gastrocnemius muscle myofiber size
Gastrocnemius Muscle COX Enzyme Activity | Measured at baseline and four-month follow up
  Four month changes in gastrocnemius muscle COX enzyme activity
Gastrocnemius Muscle Abundance of Satellite Cells | Measured at baseline and four-month follow up
  Four month changes in gastrocnemius muscle abundance of satellite cells
Gastrocnemius Muscle Abundance of Myofibers with Central Nuclei | Measured at baseline and four-month follow up
  Four month changes in gastrocnemius muscle abundance of myofibers with central nuclei
Walking Impairment Questionnaire (WIQ) Speed Score | Baseline and four-month follow-up
  Four month changes in the WIQ speed score (0-100 score, 100-best)
Walking Impairment Questionnaire (WIQ) Stair Climbing Score | Baseline and four month follow-up
  Four month changes in WIQ stair climbing score (0-100 score, 100-best).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois